CLINICAL TRIAL: NCT02976376
Title: The Box: Using Smart Technology to Improve One-year Outcome of Myocardial Infarction Patients
Acronym: TheBox
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, RoderickTreskes, BSc, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P16.070
Record Dates: First submitted 2016-08-09; First posted 2016-11-29 (Estimated); Last update posted 2018-12-06 (Actual); Status verified 2018-12

CONDITIONS: Myocardial Infarction
Keywords: Myocardial infarction; e-Health; mHealth; mobile phones; smartphone; follow-up
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- The Box (Experimental): After randomization, patients in the intervention group will receive a box ("The Box") with all the devices described above. Instructions about the installation and usage of the devices will be given. Patients will be asked to measure their weight and blood pressure once a day. Furthermore, patients will be asked to record an ECG using the AliveCor once a day. Moreover, they are asked to record an ECG in case of any symptoms of possible cardiac origin, as judged by the patient. All data will be automatically transferred to the Leiden University Medical Center. Lastly, two of the four outpatient clinical visits will be done via a video connection. The content of the interview will be comparable to the content of a regular outpatient clinic visit.
  Interventions: Other: The Box
- Control (No Intervention): Patients who are randomized to the control group will receive regular care.

INTERVENTIONS:
Other: The Box — The Box contains four smartphone compatible devices. Patients will measure their vital signs and automatically send them to the hospital.
  Arms: The Box

SUMMARY:
Study to investigate whether a smart technology intervention can improve clinical and cost-effectiveness of one-year follow-up in patients who suffered from acute myocardial infarction.

DETAILED DESCRIPTION:
Rationale: Smart technology could improve quality of care in patients after acute myocardial infarction (AMI) with either ST or non-ST elevation.

Objective: The objective of this study is to measure the effect of a smart technology intervention on patients after AMI.

Study design: The design of the study is a single-center, open randomized-controlled trial.

Study population: The study population consists of patients who have been discharged from the ward of the cardiology department of the Leiden University Medical Center after primary percutaneous coronary intervention (PCI) for either ST or non-ST elevation myocardial infarction.

Intervention: Patients will be randomized to either "The Box" or regular follow-up. Patients who have been randomized to The Box will receive a box containing a smartphone compatible electrocardiogram (ECG) monitor, a weight scale, an activity tracker and a blood pressure monitor. If patients are randomized to The Box, two of the four outpatient clinic visits will be replaced by an e-consult, in which a patient does not have to go to the hospital, but talks with his or her doctor or nurse practitioner via a secured video connection.

Main study parameters/endpoints: The primary endpoint of the study will be the percentage of patients with controlled blood pressure in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Patient is admitted with acute myocardial infarction
* Patient is able to communicate in English or Dutch at B1 level

Exclusion Criteria:

* Body Mass Index > 35 kg x m-2
* Included in another randomized controlled trial
* Patient is <18 years of age
* Patient is considered an incapacitated adult
* Patient is pregnant
* Patient is unwilling to sign the informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-05-12 (Actual); Primary Completion 2018-11-09 (Actual); Study Completion 2018-11-09 (Actual)

PRIMARY OUTCOMES:
Controlled Blood pressure | One year
  A blood pressure is considered controlled if the average of three measurements is below 140 (systolic) and 90 (diastolic) after 12 months of follow-up

SECONDARY OUTCOMES:
Patient satisfaction of received care | One year
  Patient satisfaction, defined as the hight of scores derived from validated patient satisfaction questionnaire, will be measured in both groups.
Major adverse cardiac events | One year
  Defined as cardiovascular death, recurrent STEMI, recurrent NST-ACS, revascularization, hospitalization for heart failure, TIA or ischaemic stroke
Medication-adherence | One year
  Medication adherence is measured by validated medication adherence questionnaires. This questionnaires asks if patients take their medicines in accordance to doctors advice.
Physical activity | One year
  Measured by the iPAQ questionnaire
Quality of life | One year
  Measured by the validated SF-36 questionnaire
Healthcare utilization | One year
  Defined as the number of hospital visits, defined as an outpatient clinic visit, emergency care visit or admission for any reason. This will be measured via questionnaires and verified by EMR data
Percentage of patients in which a previously unknown sustained arrhythmia (30 seconds or more) is detected | One year

CONTACTS AND LOCATIONS:
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Treskes RW, van den Akker-van Marle ME, van Winden L, van Keulen N, van der Velde ET, Beeres S, Atsma D, Schalij MJ. The Box-eHealth in the Outpatient Clinic Follow-up of Patients With Acute Myocardial Infarction: Cost-Utility Analysis. J Med Internet Res. 2022 Apr 25;24(4):e30236. doi: 10.2196/30236. PMID 35468091
- [Derived] Treskes RW, van Winden LAM, van Keulen N, van der Velde ET, Beeres SLMA, Atsma DE, Schalij MJ. Effect of Smartphone-Enabled Health Monitoring Devices vs Regular Follow-up on Blood Pressure Control Among Patients After Myocardial Infarction: A Randomized Clinical Trial. JAMA Netw Open. 2020 Apr 1;3(4):e202165. doi: 10.1001/jamanetworkopen.2020.2165. PMID 32297946
- [Derived] Treskes RW, van Winden LA, van Keulen N, Atsma DE, van der Velde ET, van den Akker-van Marle E, Mertens B, Schalij MJ. Using Smart Technology to Improve Outcomes in Myocardial Infarction Patients: Rationale and Design of a Protocol for a Randomized Controlled Trial, The Box. JMIR Res Protoc. 2017 Sep 22;6(9):e186. doi: 10.2196/resprot.8038. PMID 28939546